CLINICAL TRIAL: NCT03019250
Title: Effects of Colostrum Supplement on Inflammatory and Growth Factors, Immune System Function and Clinical Outcomes in Hospitalized Patients With Enteral Feeding in Intensive Care Unit
Brief Title: A Trial of Enteral Colostrum on Clinical Outcomes in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Ghazaleh Eslamian, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016670
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Critical Illness; Infection Complication; Multiple Organ Dysfunction Syndrome
Keywords: Colostrum; Critical Care Outcomes; Intensive Care Unit; Inflammation; Infection; mortality
MeSH Terms: conditions — Critical Illness; Multiple Organ Failure; Inflammation; Infections | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colostrum (Experimental): Intervention patients will be received enteral formula and colostrum powder 20 g/kg/day given via nasogastric tube as boluses q 4hrs.
  Interventions: Dietary Supplement: Colostrum
- Maltodextrin (Placebo Comparator): Control patients will be received enteral formula and maltodextrin mixed in with water and given via nasogastric tube as boluses q 4hrs.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Colostrum — Enteral colostrum 20g/day powdered colostrum to be mixed in with water and given via nasogastric tube q4 hrs.
  Other Names: Bovine Colostrum
  Arms: Colostrum
Dietary Supplement: Maltodextrin — Maltodextrin mixed with water given via NG tube Q 4 hours.
  Arms: Maltodextrin

SUMMARY:
Enteral administration of immune-modulating nutrients such as glutamine, omega-3 fatty acids, selenium, and antioxidants has been suggested to reduce infections and improve recovery from critical illness. However, the effects of colostrum on clinical outcomes in critical ill patients has not been investigated. In current trial, intensive care unit patients with enteral feeding will receive either enteral colostrum or maltodextrin as placebo.

DETAILED DESCRIPTION:
A randomized, double blind, controlled trial will be conducted in general intensive care unit (ICU) in Tehran, Iran. After a full review of the inclusion and exclusion criteria and explanation of the risks and benefits of the study, written consent form will be completed. Intervention patients will be received 20 g/day of colostrum along with enteral formula and control patients will be received maltodextrin along with enteral formula. Patients will be assessed for occurrence of new infection, organ failure, duration of stay in ICU, 28 days and 6 months mortality and inflammatory and immune markers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) admitted to ICU
* Start of study intervention within 48 hours after ICU admission
* Expected to require enteral nutrition for at least 72 hours aiming for full enteral nutrition and receive at least 80 percent of enteral formula during the first 48 hour
* Written informed consent of patient or written informed consent of legal representative

Exclusion Criteria:

* Enrollment in a related ICU interventional study
* Requiring other specific enteral nutrition for medical reason
* Death or Discharge before 5th day
* Having any contra-indication to receive enteral nutrition
* Pregnant patients or lactating with the intent to breastfeed
* BMI <18 or > 40.0 kg/m2
* Have life expectancy of <6 mo
* Patients who are moribund
* History of allergy or intolerance to the study product components
* Receiving colostrum during two weeks before start study product
* Have other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of infection | Day 28

SECONDARY OUTCOMES:
28-day Mortality | Day 28
6-month mortality | month 6
Length of stay in ICU | Day 28
Serum Immunity Markers | baseline, Day 5, Day 10
Serum Inflammatory Markers | baseline, Day 5, Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Ghazaleh Eslamian, MS,PhDcandid, Principal Investigator — National Nutrition and Food Technology Research Institute Shahid Beheshti University of Medical Sciences, Tehran, Iran
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim JW, Jeon WK, Kim EJ. Combined effects of bovine colostrum and glutamine in diclofenac-induced bacterial translocation in rat. Clin Nutr. 2005 Oct;24(5):785-93. doi: 10.1016/j.clnu.2005.04.004. PMID 15919136
- [Background] Rathe M, Muller K, Sangild PT, Husby S. Clinical applications of bovine colostrum therapy: a systematic review. Nutr Rev. 2014 Apr;72(4):237-54. doi: 10.1111/nure.12089. Epub 2014 Feb 26. PMID 24571383
- [Background] Benson KF, Carter SG, Patterson KM, Patel D, Jensen GS. A novel extract from bovine colostrum whey supports anti-bacterial and anti-viral innate immune functions in vitro and in vivo: I. Enhanced immune activity in vitro translates to improved microbial clearance in animal infection models. Prev Med. 2012 May;54 Suppl:S116-23. doi: 10.1016/j.ypmed.2011.12.023. Epub 2011 Dec 28. PMID 22227281